CLINICAL TRIAL: NCT06487065
Title: Observational Retrospective Study To Characterize and Assess Clinical Outcomes of Patients Receiving Tezepelumab in the Framework Of Use in Special Situations Prior to Commercialisation in Spain
Acronym: T-ROSS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00028
Record Dates: First submitted 2024-05-23; First posted 2024-07-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The aim of this study is to provide the first results on the use of tezepelumab under clinical practice conditions in severe asthma patients who participated in the "foreign medication supply" program in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 12 years and older with severe asthma who were inadequately controlled with high dose inhaled corticosteroids plus another medicinal product
* Received at least one dose of tezepelumab under the FMS program, established according to Royal Decree 1015 / 2009 (prior to commercialization)

Exclusion Criteria:

* Subjects having received tezepelumab or any other biologic for the treatment of asthma in the context of a clinical trial at any time during the 12 months prior to the index date.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of all the subjects ≥ 12 years old who have received tezepelumab in the "Foreign medication supply" (FMS) program in Spain. However, some patients may have received tezepelumab under "Foreign medication supply" program as well as marketed tezepelumab, but all of them started while FMS program was in place
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Comorbidities (e.g., allergic rhinitis, nasal polyposis, gastroesophageal reflux, chronic obstructive pulmonary disease (COPD), atopic dermatitis and other eosinophilic conditions, conditions related to OCS chronic use, etc.) | 12 months before index date and index date (date of treatment initiation with tezepelumab)
Number of respiratory infections and diseases in the previous 12 months and index date | In the previous 12 months and index date (date of treatment initiation with tezepelumab)
Exacerbations in the previous 12 months and Exacerbations from index date until all available follow-up (number and dates for each exacerbation episode) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
When available, lung function measurements including spirometry, Inspiratory Capacity, and bronchodilator reversibility test. | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  Lung function measurements including spirometry (FEV1(L), FVC(L), PEF(L/s), FEF25-75%(L/s), Inspiratory Capacity (IC) (L)), and bronchodilator reversibility test. From the spirometry measurements, the following will be calculated: FEV1/FVC ratio (%) and FEV1 % predicted (%)
Blood Eosinophil count (109 /L, mm3 ) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
IgE (IU/mL; kU/mL; ng/mL (mg/L); ng/dL (ng/100mL); ng%) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
FeNO (ppb) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
Allergy status (Prick test, RAST or similar, clinical relevance of allergy, etc.) (only baseline) | Only on the baseline (12 months prior to Index date)
Neutrophil count (10 9 /L, mm3 ) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
Sputum biomarkers: sputum eosinophils (%); sputum neutrophils (%) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
Socio-demographic variables: Age (years), Gender (male, female, other); Smoking status (Current smoker, Ex-smoker, Non-smoker) and cumulative index (packs/year); Height (cm) and weight (kg); Body Mass Index (BMI) (kg/m 2 ) | Only on the index date (If no information referred to index date is available, latest available data before the index date)
  To describe the demographic characteristics of patients

SECONDARY OUTCOMES:
Asthma Control Test (ACT) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  A short, simple, patient-based tool for identifying subjects with poorly controlled asthma. ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well controlled asthma. We will use the Spanish validation
Asthma Impairment and Risk Questionnaire (AIRQ) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  The AIRQ® is a patient assessment tool intended to help identify patients 12 years of age and older whose health may be at risk because of uncontrolled asthma. AIRQ® is a 10-item, equally weighted, yes/no composite asthma control questionnaire that includes 7 impairment and 3 risk items. AIRQ® was validated against a standard of ACT™. The combination of selected AIRQ® items and cut points of control demonstrated a sensitivity of 0.90 to identify patients whose asthma was well-controlled (cut point of ≥2), and a specificity of 0.96 to determine patients whose asthma was very poorly controlled (cut point of ≥5)
Asthma Quality of Life Questionnaire (AQLQ) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  A disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease. It is a validated, 32-question, with 2-week recall, self-administered instrument where questions are grouped into four domains: activity limitations (12 items), symptoms (11 items), emotional functions (5 items) and environmental stimuli (4 items). The questions are scored on a scale of 1-7, with higher scores indicating better quality of life
MiniAQLQ | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  This instrument has 15 questions in the same domains as the original AQLQ and takes 3-4 minutes to complete. The MiniAQLQ has very good reliability, cross-sectional validity, responsiveness and longitudinal validity. Like the AQLQ, a change in score of greater than 0.5 can be considered clinically important

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Research Site, Alcázar de San Juan
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Bilbao
  - Research Site, Coslada
  - Research Site, Donostia / San Sebastian
  - Research Site, Fuenlabrada
  - Research Site, Gran Canaria
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Talavera de la Reina
  - Research Site, Torrejón de Ardoz
  - Research Site, Valencia

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180R00028&attachmentIdentifier=df34697c-e4bb-4bd8-b0ef-5333efd8c21c&fileName=D5180R00028_CSR_Synopsis.pdf&versionIdentifier=